CLINICAL TRIAL: NCT06561620
Title: A Prospective Study of Befotertinib Adjuvant Therapy in Patients With Postoperative MRD-positive Non-small Cell Lung Cancer in Stage IA2-IB With High Risk Factors
Brief Title: Befotertinib Adjuvant Therapy in Stage IA2-IB NSCLC Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Chief of the MDT board of thoracic cancer, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ECTOP-1024
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: 3-year Disease-free Survival

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Active Comparator)
  Interventions: Drug: Befotertinib
- Observation (No Intervention)

INTERVENTIONS:
Drug: Befotertinib — Befotertinib is a novel, selective oral third-generation epidermal growth factor receptor tyrosine-kinase inhibitor.
  Arms: Treatment

SUMMARY:
To evaluate 3-year disease-free survival after complete resection in patients with MRD-positive EGFR-sensitive mutations in Stage IA2-IB NSCLC treated with adjuvant befortinib and under routine observation (3y-DFS).

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years old.
2. Gender: both men and women are acceptable, as balanced as possible.
3. Patients with lung adenocarcinoma who underwent R0 resection and were clinically confirmed as IA2-IB by histopathology and whose tumor size was (1-4cm), the surgical tissue samples tested positive for EGFR-sensitive mutations and positive for MRD after surgery.
4. Accompanied by arbitrary ≥ 2 high-risk factors; High risk factors such as pleural invasion, airway diffusion, vascular infiltration, low differentiation, pathological micropapillary composition ≥ 15%, complex glandular composition ≥ 20%, etc.

4. Achieve R0 resection: For CTR < 50% ground glass nodules, wedge resection is acceptable and the margin is negative, and 3 groups of lymph node biopsies are negative; for CTR ≥ 50% or pure solid nodules, at least segmental resection is undergone, and lymph node dissection is systematically performed; if there is no clear evidence of metastasis, if it cannot be judged, it can be determined by an independent review committee for pathological consultation.

5. The ECOG behavioral status score is 0 to 1, and the expected survival time is > 1 year.

6. Voluntary MRD screening and voluntary befortinib adjuvant therapy; 7. Have a certain organ system function, defined as follows, based on the researcher's experience A. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L B. Platelets ≥ 100 x 109/L; C. Hemoglobin ≥ 9 g/dL (≥ 90 g/L) Note that in order to achieve the required hemoglobin level, blood transfusion is allowed; D. Total bilirubin ≤ 1.5 times the upper limit of normal (ULN); E. If there is no liver metastasis, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; if liver metastasis, ≤ 5 × ULN; F. Creatinine ≤ 1.5 x ULN. Patients are still eligible for inclusion if the creatinine clearance value calculated by the Cockcroft-Gault method is ≥ 50 mL/min (0.83 mL/s).

8. Female subjects of childbearing age must have a serum pregnancy test within 3 days before the start of the study drug, and the result is negative, and they are willing to use a medically approved high-efficacy contraceptive method (such as intrauterine devices, contraceptives or condoms) during the study period and within 3 months after the last administration of the study drug; for significant other male subjects who are women of childbearing age, they should be surgically sterilized, or agree to use effective methods of contraception during the study period and within 3 months after the last study dose.

9. Voluntary and capable of following the test and follow-up procedures. 10. Sign the informed consent form.

Exclusion Criteria:

1. There is any other treatment before the operation, and no informed consent is signed;
2. The patient has been diagnosed with cancer within 2 years;
3. Have a history of interstitial lung disease, drug-induced interstitial disease or any active interstitial lung disease with clinical evidence; CT scan at baseline revealed idiopathic pulmonary fibrosis.
4. Patients who are known to be allergic to any component of befortinib or similar drugs;
5. Pregnant or lactating women;
6. Situations considered unsuitable for inclusion by other researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2029-05-01 (Estimated)

PRIMARY OUTCOMES:
3-year disease-free survival | 3 years
  3-year disease-free survival after complete resection in patients with MRD-positive EGFR-sensitive mutations in Stage IA2-IB NSCLC

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No